CLINICAL TRIAL: NCT02051400
Title: Evaluation of McGrath® MAC Using Glidescope® Ranger for Novice Providers in a Simulated Difficult Airway: A Randomised Manikin Study
Brief Title: Evaluation of McGrath® MAC Video Laryngoscope
Acronym: EMMVL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Wonhee Kim, Emergency Medicine Fellow, Department of Emergency Medicine, Hanyang University Seoul Hospital, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: McGrath® MAC 1
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Intubation; Difficult
Keywords: Intubation; Laryngoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intubation with the McGrath® MAC video laryngoscope (Experimental): Participants perform five intubation attempts using the airway manikin with the normal airway setting. After completing the normal airway session, the participants performed another five attempts with the neck immobilization setting using a neck collar.
  Interventions: Device: the McGrath® MAC video laryngoscope; Device: the GlidesScope® Ranger video laryngoscope; Device: the Macintosh laryngoscope
- Intubation with the GlidesScope® Ranger video laryngoscope (Experimental): Participants perform five intubation attempts using the airway manikin with the normal airway setting. After completing the normal airway session, the participants performed another five attempts with the neck immobilization setting using a neck collar.
  Interventions: Device: the McGrath® MAC video laryngoscope; Device: the GlidesScope® Ranger video laryngoscope; Device: the Macintosh laryngoscope
- Intubation with Macintosh laryngoscope (Experimental): Participants perform five intubation attempts using the airway manikin with the normal airway setting. After completing the normal airway session, the participants performed another five attempts with the neck immobilization setting using a neck collar.
  Interventions: Device: the McGrath® MAC video laryngoscope; Device: the GlidesScope® Ranger video laryngoscope; Device: the Macintosh laryngoscope

INTERVENTIONS:
Device: the McGrath® MAC video laryngoscope
Device: the GlidesScope® Ranger video laryngoscope
Device: the Macintosh laryngoscope

SUMMARY:
The purpose of this study is to evaluate whether the McGrath® MAC video laryngoscope is equal or superior when compared to the Glidescope® Ranger and the Macintosh laryngoscope for novice users in a simulated airway manikin.

DETAILED DESCRIPTION:
Investigators compared two portable video laryngoscopes (the GlidesScope® Ranger (Verathon Inc, Bothell, WA, USA) and the McGrath® MAC (Aircraft Medical Ltd, Edinburgh, UK)) and a German type Macintosh metal blade with a fiberoptic light. A blade size of 4 was used on all devices. All intubations using video laryngoscopes were performed according to the manufacturers' instructions. A specialised rigid stylet (the GlideRite®) was used with the Glidescope® and a flexible plastic stylet bent with a hockey stick curvature, was used with the McGrath® MAC and the Macintosh laryngoscope. A size 7.5 endotracheal tube (Mallinckrodt™ Hi-Lo Oral/Nasal Tracheal Tube Cuffed Murphy Eye, Covidien, Ireland) was used with all the laryngoscopes.

All participants were randomly divided into 3 device groups. Each group was allowed to attempt to perform endotracheal intubation five more times using the Laerdal® Airway Management Trainer (Laerdal Medical Korea Ltd., Seoul, Korea) with the normal airway setting. After completing the normal airway session, the participants performed another five attempts with the neck immobilisation setting using a neck collar.

The sequence in which the three devices were used was randomly assigned, and all participants performed the same sequence at intervals of five weeks during the study.

ELIGIBILITY:
Inclusion Criteria:

* Medical students without previous experience of intubation

Exclusion Criteria:

* Heart, wrist, or low back disease or who were pregnant were excluded

Ages: 22 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Intubation parameter | 1st intubation attempt, an expected average of 1 min
  1. The rate for successful intubation
  2. Time to intubation
  3. The Cormack-Lehane grade at laryngoscopy
Intubation parameter | 2nd intubation attempt, an expected average of 1 min
  1. The rate for successful intubation
  2. Time to intubation
  3. The Cormack-Lehane grade at laryngoscopy
Intubation parameter | 3rd intubation attempt, an expected average of 1 min
  1. The rate for successful intubation
  2. Time to intubation
  3. The Cormack-Lehane grade at laryngoscopy
Intubation parameter | 4th intubation attempt, an expected average of 1 min
  1. The rate for successful intubation
  2. Time to intubation
  3. The Cormack-Lehane grade at laryngoscopy
Intubation parameter | 5th intubation attempt, an expected average of 1 min
  1. The rate for successful intubation
  2. Time to intubation
  3. The Cormack-Lehane grade at laryngoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk Joong Choi, MD, PhD, Study Director — Hanyang University
Locations (1):
- Hanyang University Guri Hospital, Guri-si, Kyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim W, Choi HJ, Lim T, Kang BS. Can the new McGrath laryngoscope rival the GlideScope Ranger portable video laryngoscope? A randomized manikin study. Am J Emerg Med. 2014 Oct;32(10):1225-9. doi: 10.1016/j.ajem.2014.07.034. Epub 2014 Aug 2. PMID 25171799